CLINICAL TRIAL: NCT02912533
Title: A Long-term Study of JR-131 in Renal Anemia Patients With Chronic Kidney Disease (CKD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Collaborators: JCR Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Masking: None
Other Study IDs: JR-131-302
Record Dates: First submitted 2016-09-21; First posted 2016-09-23 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

ARMS (1):
- JR-131 (Experimental)
  Interventions: Drug: JR-131

INTERVENTIONS:
Drug: JR-131

SUMMARY:
The purpose of this study is to investigate the safety and efficacy for 52-week dosing of JR-131 in renal anemia patients with chronic kidney disease (CKD).

ELIGIBILITY:
Inclusion Criteria:

* Patients being treated with erythropoiesis stimulating agent.

Exclusion Criteria:

* Patients having complication or history of a cardiovascular / lung / brain infarction.
* Patients having a pronounced hemorrhagic lesion.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2016-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Measure adverse events | 52 weeks

SECONDARY OUTCOMES:
Hemoglobin level | 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple Locations, Japan